CLINICAL TRIAL: NCT01458353
Title: Microbiological Spectrum of the Intraperitoneal Surface After Elective Right-sided Colon Cancer: Are There Differences in the Peritoneal Contamination After Performing a Stapled or a Handsewn Anastomosis?
Brief Title: Microbiological Spectrum of the Intraperitoneal Surface After Elective Right-sided Colon Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Doctor in Surgery by Universidad Autonoma de Madrid (Spain), Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HGUElche1
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Peritoneal Contamination After Ileocolonic Anastomosis; Wound Infection; Intra-abdominal Abscess
Keywords: Right-sided colon cancer; Ileocolonic anastomosis; stapled anastomosis; handsewn anastomosis; peritoneal contamination; microbiological spectrum
MeSH Terms: conditions — Wound Infection; Abdominal Abscess

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Handsewn ileocolonic anastomosis (Experimental): Swabs obtained from patients undergoing handsewn ileocolonic anastomosis
  Interventions: Procedure: Handsewn anastomosis
- Stapled ileocolonic anastomosis (Experimental): Swabs obtained for culture in those patients undergoing stapled ileocolonic anastomosis
  Interventions: Procedure: Stapled anastomosis

INTERVENTIONS:
Procedure: Stapled anastomosis — Stapled anastomosis after ileocolonic resection
  Arms: Stapled ileocolonic anastomosis
Procedure: Handsewn anastomosis — Handsewn anastomosis after ileocolonic resection
  Arms: Handsewn ileocolonic anastomosis

SUMMARY:
Despite performing colonic surgery with strict asepsia measures, minimizing the contact of the colon lumen with the peritoneum, some contamination is nearly impossible to avoid. In stapled anastomosis, the hole opened in the colon is minimum, just the necessary for introducing the parts of the mechanical devices. In handsewn anastomosis, the colonic lumen is more exposed to the peritoneum, despite the colonic occlusion with clamps meanwhile the suture is performed.

Hypothesis: After stapled anastomoses, the peritoneal contamination should be lower than after handsewn ones.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of right-sided colon cancer and plans to undergo an elective surgery with curative aims.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Peritoneal contamination after finishing the ileocolonic anastomosis | 1 year
  Swabs will be obtained from the peritoneal surface for microbiological culture

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, MD, PhD, Principal Investigator — Hospital General de Elche; Antonio Arroyo, MD, PhD, Study Director — Hospital General de Elche
Locations (1):
- Hospital General de Elche, Elche, Alicante, Spain

REFERENCES:
- [Derived] Ruiz-Tovar J, Santos J, Arroyo A, Llavero C, Lopez A, Frangi A, Armananzas L, Alcaide MJ, Candela F, Calpena R. Microbiological spectrum of the intraperitoneal surface after elective right-sided colon cancer: are there differences in the peritoneal contamination after performing a stapled or a handsewn anastomosis? Int J Colorectal Dis. 2012 Nov;27(11):1515-9. doi: 10.1007/s00384-012-1492-9. Epub 2012 May 12. PMID 22581209